CLINICAL TRIAL: NCT01317160
Title: Intermittent Pneumatic Compression Effects on Venous Thromboembolism Incidence and Healing of Achilles Tendon Rupture
Brief Title: Compression Treatment Effects on Complications and Healing of Achilles Tendon Rupture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Region Stockholm (Other Government); DJO Incorporated (Industry)
Responsible Party: Principal Investigator, Paul Ackermann, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPC-Achilles; SLL20100168 (Other Grant/Funding Number: ALF - Stockholm County Council and Karolinska Institutet)
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Rupture; Venous Thromboembolism; Venous Thrombosis; Surgical Wound Infection
Keywords: Achilles Tendon; Immobilization; Wound Healing; Intermittent Pneumatic Compression; Ultrasonography; Microdialysis
MeSH Terms: conditions — Rupture; Venous Thromboembolism; Venous Thrombosis; Surgical Wound Infection | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine care: Plaster Cast Treatment (No Intervention): Two weeks of postoperative conventional lower limb plaster cast immobilization in 30 degrees of plantarflexion
- Intermittent pneumatic compression (IPC) (Experimental): Two weeks of calf IPC by Aircast® VenaFlow® Elite System during immobilization in an orthosis Aicast® XP Walker.
  Interventions: Device: Intermittent pneumatic compression (IPC)

INTERVENTIONS:
Device: Intermittent pneumatic compression (IPC) — 6 hours IPC, daily, applied to both calves during two weeks post-operatively. The VenaFlow Elite system (Aircast, Vista, California) uses calf cuffs containing two overlapping air chambers located posteriorly on the leg. As the device cycles, the distal chamber inflates to 52 mm Hg over half a second. During the last 0.2 second of this period, the proximal chamber inflates and reaches 45 mm Hg. After six seconds of inflation the cuff deflates, and the cycle is repeated every minute.
  Other Names: VenaFlow Elite system; VenaFlow® System
  Arms: Intermittent pneumatic compression (IPC)

SUMMARY:
This prospective randomized study aims to determine whether intermittent pneumatic compression (IPC), 75 patients, beneath functional bracing compared to treatment-as-usual in plaster cast, 75 patients, can reduce the Venous Thromboembolism (VTE) incidence and promote healing of sutured acute Achilles tendon ruptures.

At two weeks post surgery, the IPC intervention will be ended and both patient groups will be immobilized in an orthosis until follow-up at six weeks.

The endpoint of the first part of the study is VTE events. The primary outcome will be the DVT-incidence at two weeks, assessed using screening compression duplex ultrasound (CDU) by two ultrasonographers masked to the treatment allocation. Secondary outcome will be the DVT-incidence at 6 weeks.

1) Deep Vein Thrombosis (DVT) detected by CDU , 2) isolated calf muscle vein thrombosis (ICMVT) detected by CDU, 3) symptomatic DVT or ICMVT detected by CDU, 4) symptomatic pulmonary embolism detected by computer tomography.

The endpoint of the second part of the study is tendon healing quantified at 2 weeks by microdialysis followed by quantification of markers for tendon repair.

The endpoint of the third part of the study is the functional outcome of the patients at one year post-operatively using four reliable and valid scores, i.e. the Achilles tendon Total Rupture Score (ATRS), Physical Activity scale (PAS), Foot and Ankle Outcome Score (FAOS) and EuroQol Group's questionnaire (EQ-5D) as well as the validated heel-rise test.

DETAILED DESCRIPTION:
The incidence of DVT after Achilles tendon rupture is as high as 30-40% and patients exhibit a prolonged healing process with variable outcome. Moreover, it has been demonstrated that low molecular weight heparin had no effect on preventing DVT after Achilles tendon surgery. Whether intermittent pneumatic compression (IPC) can prevent DVTs and improve healing after Achilles tendon rupture has to our knowledge not been tested before.

ELIGIBILITY:
Inclusion Criteria:

* Achilles tendon rupture operated on within 96 hours of diagnose.

Exclusion Criteria:

1. Inability or refusal to give informed consent for participation in the study
2. Ongoing treatment with anticoagulant therapy
3. Inability to comply with the study instructions
4. Known kidney disorder
5. Heart failure with pitting oedema
6. Thrombophlebitis
7. Recent thromboembolic event (during the preceding 3 months)
8. Recent surgery (during the preceding month)
9. Presence of known malignancy
10. Current bleeding disorder
11. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2015-08 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul W Ackermann, MD, PhD, Principal Investigator — Karolinska University Hospital, 171 76 Stockholm, SWEDEN
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Plan to share data on primary outcome (DVT)
Supporting Information: Study Protocol, SAP
Time Frame: Starting 12 months after publication the data will be available for 10 years after the study is published.
Access Criteria: Contact PI.

REFERENCES:
- [Result] Domeij-Arverud E, Labruto F, Latifi A, Nilsson G, Edman G, Ackermann PW. Intermittent pneumatic compression reduces the risk of deep vein thrombosis during post-operative lower limb immobilisation: a prospective randomised trial of acute ruptures of the Achilles tendon. Bone Joint J. 2015 May;97-B(5):675-80. doi: 10.1302/0301-620X.97B5.34581. PMID 25922463
- [Result] Abdul Alim M, Domeij-Arverud E, Nilsson G, Edman G, Ackermann PW. Achilles tendon rupture healing is enhanced by intermittent pneumatic compression upregulating collagen type I synthesis. Knee Surg Sports Traumatol Arthrosc. 2018 Jul;26(7):2021-2029. doi: 10.1007/s00167-017-4621-8. Epub 2017 Jul 1. PMID 28668970
- [Derived] Chen J, Wang J, Hart DA, Zhou Z, Ackermann PW, Ahmed AS. Complement factor D regulates collagen type I expression and fibroblast migration to enhance human tendon repair and healing outcomes. Front Immunol. 2023 Sep 6;14:1225957. doi: 10.3389/fimmu.2023.1225957. eCollection 2023. PMID 37744351
- [Derived] Wu X, Chen J, Sun W, Hart DA, Ackermann PW, Ahmed AS. Network proteomic analysis identifies inter-alpha-trypsin inhibitor heavy chain 4 during early human Achilles tendon healing as a prognostic biomarker of good long-term outcomes. Front Immunol. 2023 Jul 6;14:1191536. doi: 10.3389/fimmu.2023.1191536. eCollection 2023. PMID 37483617
- [Derived] Chen J, Wang J, Wu X, Simon N, Svensson CI, Yuan J, Hart DA, Ahmed AS, Ackermann PW. eEF2 improves dense connective tissue repair and healing outcome by regulating cellular death, autophagy, apoptosis, proliferation and migration. Cell Mol Life Sci. 2023 Apr 21;80(5):128. doi: 10.1007/s00018-023-04776-x. PMID 37084140
- [Derived] Chen J, Wang J, Hart DA, Ahmed AS, Ackermann PW. Complement factor D as a predictor of Achilles tendon healing and long-term patient outcomes. FASEB J. 2022 Jun;36(6):e22365. doi: 10.1096/fj.202200200RR. PMID 35596679
- [Derived] Svedman S, Juthberg R, Edman G, Ackermann PW. Reduced Time to Surgery Improves Patient-Reported Outcome After Achilles Tendon Rupture. Am J Sports Med. 2018 Oct;46(12):2929-2934. doi: 10.1177/0363546518793655. Epub 2018 Aug 31. PMID 30169112
- [Derived] Alim MA, Svedman S, Edman G, Ackermann PW. Procollagen markers in microdialysate can predict patient outcome after Achilles tendon rupture. BMJ Open Sport Exerc Med. 2016 Jun 10;2(1):e000114. doi: 10.1136/bmjsem-2016-000114. eCollection 2016. PMID 27900179

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Routine Care: Plaster Cast Treatment | Intermittent Pneumatic Compression (IPC)
Started | 75 | 75
Allocation to Treatment | 74 (1 patient was incorrect included) | 74 (1 patient was incorrect included)
Completed | 71 | 69
Not Completed | 4 | 6
Not completed — Incorrect inclusion | 1 | 1
Not completed — Lost to Follow-up | 3 | 3
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Care: Plaster Cast Treatment | Intermittent Pneumatic Compression (IPC) | Total
Number analyzed (Participants) | 71 | 69 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 69 | 139
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 39.9 [18 to 71] | 40.9 [26 to 62] | 40.4 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 58 | 61 | 119
Region of Enrollment [Number; unit: participants]
  Sweden | 71 | 69 | 140
Tobacco user [Number; unit: participants]
  Tobacco user: Yes | 8 | 5 | 13
  Tobacco user: No | 63 | 64 | 127
Body mass index [Mean (Full Range); unit: Kg/m/m] | 26.7 [20.2 to 35.7] | 27.1 [21 to 41.2] | 26.9 [20.2 to 41.2]

OUTCOME MEASURES:

1. Primary Outcome: Venous Thromboembolic Events (VTE)
Description: At 2 weeks postoperatively the number of participants with VTE events will be assessed by:
  1) DVT detected by compression duplex ultrasound (CDU) , 2) isolated calf muscle vein thrombosis (ICMVT) detected by CDU, 3) symptomatic DVT or ICMVT detected by CDU, 4) symptomatic pulmonary embolism detected by computer tomography.
Time Frame: 2 weeks
Population: Non-compliance was defined by exposure to less than ten hours of IPC. Therefore, two patients were withdrawn on this basis and the treatment group comprised 67 patients at final analysis.
Measure: Number; unit: participants
Arm/Group | Routine Care: Plaster Cast Treatment | Intermittent Pneumatic Compression (IPC)
Number analyzed (Participants) | 71 | 67
participants | 26 | 14
Statistical Analysis 1: Comparison: Routine Care: Plaster Cast Treatment vs Intermittent Pneumatic Compression (IPC); Domeij-Arverud et al., Bone Joint J 2015;97-B:675-80; Test type: Superiority or Other; p = 0.042, Chi-squared
Statistical Analysis 2: Comparison: Routine Care: Plaster Cast Treatment vs Intermittent Pneumatic Compression (IPC); Test type: Superiority or Other; p < 0.05, Regression, Logistic; Age was adjusted for in the calculation; Odds Ratio (OR) = 2.81, 95% CI 2-sided [1.25 to 6.32] — Risk of VTE by routine care (numerator) divided by IPC treatment (denominator)

2. Secondary Outcome: Functional Outcome - Muscular Endurance Tests (Heel-rise)
Description: The functional outcome was assessed at 1year post-operatively by the validated calf muscle endurance test, i.e. heel rise test (Silbernagel KG et al. A new measurement of heel-rise endurance with the ability to detect functional deficits in patients with Achilles tendon rupture. Knee Surg Sports Traumatol Arthrosc. 2010). The Muscle lab linear encoder (Ergotest Technology, Oslo, Norway), was used for data collection. Standardized footwear was used. Patients warmed up before testing. During the heel-rise test, verbal encouragement was used. The patient was instructed to go as high as possible on each heel-rise with a straight knee. A metronome was used for standardized frequency of 30 heel-rises per minute. The test was terminated when the patient stopped or could not maintain frequency. For analysis, the limb symmetry index (LSI, percentage of injured vs. uninjured side) values were used.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: Index of Injured versus uninjured side
Arm/Group | Routine Care: Plaster Cast Treatment | Intermittent Pneumatic Compression (IPC)
Number analyzed (Participants) | 70 | 56
Index of Injured versus uninjured side
  LSI of average height of heel-rise | 78.5 (14.6) | 82.5 (17.0)
  LSI of Eccentric power (W) | 78.2 (15.8) | 82.6 (22.9)
  LSI of Heel-rise repetitions | 83.0 (22.5) | 84.1 (19.1)
  LSI of total concentric work (J) | 66.8 (22.2) | 69.4 (20.1)
  LSI of concentric power (W) | 81.3 (24.3) | 74.2 (32.3)

3. Secondary Outcome: Venous Thromboembolic Events (VTE)
Description: At 6 weeks postoperatively the number of participants with VTE events will be assessed by:
  1) DVT detected by compression duplex ultrasound (CDU) , 2) isolated calf muscle vein thrombosis (ICMVT) detected by CDU, 3) symptomatic DVT or ICMVT detected by CDU, 4) symptomatic pulmonary embolism detected by computer tomography.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Routine Care: Plaster Cast Treatment | Intermittent Pneumatic Compression (IPC)
Number analyzed (Participants) | 71 | 69
participants | 34 | 36
Statistical Analysis 1: Comparison: Routine Care: Plaster Cast Treatment vs Intermittent Pneumatic Compression (IPC); Test type: Superiority or Other; p = 0.737, Chi-squared

4. Secondary Outcome: Patient-reported Outcome
Description: The patients' symptoms will be assessed using the Achilles tendon Total Rupture Score (0-100, 100=best)
Time Frame: One year
Population: Achilles tendon Total Rupture Score (0-100, 100=best outcome) is presented here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Routine Care: Plaster Cast Treatment | Intermittent Pneumatic Compression (IPC)
Number analyzed (Participants) | 64 | 55
score on a scale | 78 (19.3) | 77.8 (17.2)

5. Secondary Outcome: Microdialysis
Description: At 2 weeks postoperatively in-vivo microdialysis will be performed on as described by Greve et al 2012 (DOI: 10.1111/j.1600-0838.2012.01475.x).
  In the microdialysate substances will be assessed, eg. markers of tendon callus production, procollagen type I (PINP), by enzymatic quantification.
Time Frame: 2 weeks
Population: Concentration of procollagen type I (PINP) ng/ml.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Routine Care: Plaster Cast Treatment | Intermittent Pneumatic Compression (IPC)
Number analyzed (Participants) | 19 | 14
ng/mL | 2.05 (0.78) | 3.47 (1.81)

6. Secondary Outcome: Time From Injury to Surgery
Description: Prognostic factor:
  Time to surgery , i.e. the time from ATR injury to start of the surgical procedure, will be calculated by using the time-point at which the patient sustained the injury as described in the patient journal, as well as the starting time point of the surgery as registered in the computerized operation report.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Routine Care: Plaster Cast Treatment | Intermittent Pneumatic Compression (IPC)
Number analyzed (Participants) | 70 | 69
hours | 62.33 (24.45) | 62.18 (26.19)

7. Other Pre Specified Outcome: Surgeon Sex
Description: Prognostic factor: All patients are operated on according to a standardized surgical protocol. and the surgeon on duty will perform the surgical repair and no specific surgeon can be selected by the patients. Unknown sex of the operating surgeon will be included as an additional exclusion criterion in the study.
Time Frame: Surgery will be performed within 10 days of injury
Reporting Status: Not Posted, anticipated posting 2024-08

8. Other Pre Specified Outcome: Surgeon Experience
Description: Prognostic factor: All patients are operated on according to a standardized surgical protocol. and the surgeon on duty will perform the surgical repair and no specific surgeon can be selected by the patients. The experienced group of surgeons will consist of specialists accredited with a specialist licence issued by The Swedish National Board of Health and Welfare. The less experienced group of surgeons will consist of residents.
Time Frame: Surgery will be performed within 10 days of injury
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: At outpatients visit
Arm/Group | Routine Care: Plaster Cast Treatment | Intermittent Pneumatic Compression (IPC)
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71
Other Adverse Events (participants affected / at risk) | 5/71 | 3/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Routine Care: Plaster Cast Treatment (N=71) | Intermittent Pneumatic Compression (IPC) (N=69)
Infections (Infections and infestations) | 4 (4) | 2 (2) — Local infections
Re-rupture (Surgical and medical procedures) | 1 (1) | 1 (1) — Re-rupture of the Achilles tendon occurring before the 6 weeks follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No